CLINICAL TRIAL: NCT01117883
Title: Effect of Gentle Sternal Chest Wall Pressure on Central Hemodynamic Measurements and Intrathoracic Pressure During Mechanical Ventilation in Children
Brief Title: Sternal Wall Pressure in the Cath Lab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Laerdal Foundation for Acute Care Medicine (Unknown)
Responsible Party: Andrew Galtz, MD, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-007428
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Perfusion Pressures; Central Venous Pressure; Cardiac Output; CPR; Cardiac Arrest
Keywords: Perfusion pressures; central venous pressure; cardiac output; CPR; cardiac arrest; Leaning; incomplete release
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Application of two different sternal weights — Two separate weights (first 10% of body weight, then 20% of body weight) will be placed on the sternum and changes in central hemodynamic measurements and intrathoracic pressure will be recorded and documented.

SUMMARY:
This protocol is a prospective interventional pilot study at the Children's Hospital of Philadelphia to determine whether or not two increments of sternal pressure known to occur during "leaning" in CPR affects hemodynamic function, coronary perfusion pressures, and intrathoracic pressure in order to inform the resuscitation community on reasonable target pressures to avoid "leaning" on the chest during pediatric CPR.

DETAILED DESCRIPTION:
STUDY RATIONALE The critical importance of positive and negative intrathoracic pressures during Cardiopulmonary Resuscitation (CPR) has been recently demonstrated. During CPR, excessive positive intrathoracic pressure caused by overzealous ventilation or incomplete chest wall decompression has a detrimental effect on venous return to the heart, cardiac hemodynamics, and survival in adults. FDA-approved monitor/defibrillators with sensors that detect and provide feedback on the quality of chest compressions, including the amount of sternal pressure ("leaning"), can improve the quality of CPR in adults. These monitor/defibrillators have recently been implemented in the PICU and ED at CHOP. However, determining whether "leaning" (or gentle sternal pressure) affects return of venous blood to the thorax and intrathoracic pressure in children is unknown. A pilot study to determine whether or not two increments of sternal pressure known to occur during "leaning" in CPR affects hemodynamic function, coronary perfusion pressures, and intrathoracic pressure would be a first step toward informing the resuscitation community on reasonable target pressures to avoid "leaning" on the chest during pediatric CPR.

STUDY OBJECTIVE(S)

* To characterize the effect of the application of two different weights on the sternum known to approximate "leaning" during CPR on central hemodynamic measurements and coronary perfusion pressures in mechanically ventilated children.
* To characterize the effect of the application of two different weights on the sternum known to approximate "leaning" during CPR on intrathoracic pressure in mechanically ventilated children STUDY DESIGN This protocol is a prospective interventional pilot study at the Children's Hospital of Philadelphia.

STUDY PHASES Screening: Prospective patients enrolled will be screened by a co-investigator. Those that meet inclusion criteria will be approached by a member of the investigative team during the routine pre-procedure evaluation in the Cardiac Intake Center for discussion of the study and informed consent.

Phase 1: We will measure the depth of the chest. We will measure central hemodynamic pressures and function, coronary perfusion pressures and intrathoracic pressures as two weights (10% and 20% of body weight) are placed on the sternum. The primary outcome variable will be the change in any of the central hemodynamic measurements before and after each weight is applied to the sternum.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 months to < 8 years.
2. Weight 5 to 50 kilograms.
3. Hemodynamically stable (pre-anesthetic vital signs will be within normal range of expected for age and stability during the procedure is defined as no fluctuation in heart rate or blood pressure >20%. Ultimate determination of hemodynamic stability for inclusion will be defined by the attending Anesthesiologists and Interventional Cardiologists involved in the procedure)
4. Volume Limited Ventilation Mode on Conventional Mechanical Ventilator using either cuffed or uncuffed endotracheal tubes with minimal leak (leak >30 mmHg).
5. Heart transplant recipients presenting for a routine, scheduled, surveillance cardiac catheterization per standard clinical protocol.
6. Greater than 6 months removed from date of cardiac transplant.
7. Normal cardiac function (defined as a shortening fraction of ≥ 30% or qualitatively described as "normal" if a m-mode shortening fraction was not obtained) with normal function of all valves (defined as insufficiency of all valves as either "none", "trivial", or "mild") on their pre-procedure echocardiogram.

Exclusion Criteria:

1. Patients with contraindication to gentle, direct chest wall pressure (e.g. fresh sternotomy, recent chest wall surgery or chest tube in place)
2. Patients with an implantable pacemaker or AICD.
3. Patients on beta blockers.
4. Patients not in normal sinus rhythm on their pre-procedural ECG.
5. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study procedures.
6. Non-English speaking families

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in central hemodynamic measurements with application of two different sternal weights. | 1 yr

SECONDARY OUTCOMES:
The secondary endpoint is the change in end-expiratory intrathoracic pressure with application of two different sternal weights. | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Andy Glatz, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States